CLINICAL TRIAL: NCT05812274
Title: A Phase IV Study of Apricity C.A.R.E. Program for Cancer Adverse Events Rapid Evaluation to Improve Treatment Outcomes of Ethnic/Racial Minority Non-small Cell Lung Cancer (NSCLC) Patients Receiving Immunotherapy
Brief Title: Apricity CARE to Improve ICI Outcomes of Ethnic/Racial Minority NSCLC Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Brian Henick, MD, Assistant Professor of Medicine at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAU2705
Record Dates: First submitted 2023-03-30; First posted 2023-04-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Immune-Checkpoint Inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: People who meet eligibility requirements and provide informed consent will be randomly allocated to the two arms with a 1:1 allocation ratio.The randomization will match patients according to: 1) age, 2) performance status (ECOG <2 vs >=2) and 3) receiving ICI monotherapy vs. ICI plus chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants are provided with ApricityRx digital solution with pulse oximeters and 24/7 C.A.R.E. (Cancer Adverse event Rapid Evaluation) to monitor and capture ePRO, identify onset or progression of symptoms verified by nurse triage, trigger intervention by the study team.
  Interventions: Other: Apricity C.A.R.E. Program for Cancer Adverse events Rapid Evaluation
- Control Arm (No Intervention): Clinicians will monitor NSCLC patients on ICIs for irAEs as a standard of care using routine practices.

INTERVENTIONS:
Other: Apricity C.A.R.E. Program for Cancer Adverse events Rapid Evaluation — The Apricity CARE program for Cancer Adverse events Rapid Evaluation is a cloud-based 24/7 on-demand clinical coverage service, delivered exclusively via the ApricityRx digital care platform by certified and licensed healthcare professionals who are trained to monitor patient's symptoms and conduct standardized triage following guideline-based or protocol-specified pathways with 3 parts:
  * ApricityCare™ Mobile Application - to collect health data (PGHD) on biometrics and self-reported symptoms (PRO) of symptoms and potential side effects at home, in between doctors' visits, and offers educational content in video.
  * ApricityOncology™ Web-based Application - to provide authorized healthcare providers an organized, longitudinal and summarized view of a patient's pertinent cancer history and real world PGHD for purpose of symptom monitoring.
  * ApricityManage™ Dashboard - a dashboard intended for administrators, sponsors or funders to track program status.
  Other Names: Apricity CARE program
  Arms: Intervention Arm

SUMMARY:
The purpose of this trial is to study the effectiveness of the AprictyRxTM care service to improve treatment outcomes of ethnic/racial minority N.S.C.L.C. patients receiving standard of care immunotherapy, and reduce the frequency of healthcare system interactions.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (I.C.I.) targeting the PD-1/PD-L1 axis have changed the treatment landscape of non-small cell lung cancer (N.S.C.L.C.). After demonstrating improved efficacy and tolerability compared to standard chemotherapy in several large clinical trials, these novel drugs are now F.D.A. approved in multiple treatment settings. With the increase in I.C.I. use, the incidence of immune-related adverse effects (irAEs) has also risen, occurring in up to 16% of ICI-treated patients. Prompt recognition and timely management are necessary to avert potential poor outcomes from direct toxicity and/or early treatment discontinuation. However, rapid adoption of I.C.I.s may limit healthcare providers' experience and comfort with managing important irAEs. Additionally, existing barriers to access care that disproportionately impact racial and ethnic minority patients may amplify the inability to manage patients on I.C.I.s effectively.

Using technologically-enabled health interventions in a culturally competent manner can improve access to health care resources and reduce health disparities. These platforms need to be optimized at the literacy level of underserved minority communities and can be adapted to meet the community's needs. Recently, technology-enabled services focused on patient-reported outcomes have garnered growing interest in oncology.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years
* Confirmed NSCLC diagnosis
* Prescribed treatment with immune-checkpoint inhibitor, including in combination with chemotherapy
* Ability to understand and the willingness to sign a written informed consent document
* Self-identification as a member of an ethnic minority or underserved population.

Exclusion Criteria:

* An individual with presence of any medical, psychological, or social condition that, in the opinion of the investigator would preclude participation in this study.
* Patients enrolled in other interventional clinical trials at the time of screening will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Mean Likert-type scale score | 2 years
  Two focus group discussions (FGDs), stratified on a Likert-type scale based on the frequency of utilization, to determine factors related to usage of ApricityCare app and utilization of the CARE monitoring service (Run-in phase). To assess factors related to suboptimal and optimal use of the ApricityCare app and the CARE monitoring service, collectively "the Apricity CARE program".
Percent of study patients who experienced treatment delay/discontinuation | 2 years
  To determine the impact of the the Apricity CARE program on immunotherapy toxicity monitoring for N.S.C.L.C. patients receiving immunotherapy in a highly diverse New York City community. Immune Checkpoint Inhibitor (ICI) treatment delay or discontinuation is defined as a gap between doses of ICI beyond 60 days and/or the initiation of another cancer therapy without evidence of disease progression.

SECONDARY OUTCOMES:
Percent of study patients who experience a severe irAE (grade 3 or higher). | 2.5 years
  To assess the percent of study patients who experience a severe irAE (grade 3 or higher) while on study. Information about individual treatment toxicities (i.e., type, frequency) will be obtained and recorded from the ApricityRxTM platform and patient's clinical note. Toxicity grade will be assigned using the NCI CTCAE v5.0 and tallied.
Time to irAE management | 2.5 years
  To quantify time to irAE management with ICI. This will be defined as the time from the onset of irAE to time of active intervention (i.e., change in administration schedule, new prescription of supportive medication, telephone counseling about symptoms, unscheduled visits or referrals). Information will be obtained and recorded from the ApricityRxTM platform and patient's clinical note, and tallied. Unit measured in days.
Time to treatment discontinuation with ICI | 2.5 years
  To quantify time to irAE management with ICI. This will be determined as starting date of ICI to date of the last dose of ICI for any reason specified by patient's EMR. Information will be obtained and recorded from the ApricityRxTM platform and patient's clinical note, and tallied. Unit measured in days.
Number of interactions with the care team and utilization | 2.5 years
  This will be quantified as the number of clinical interactions between patients and providers from the patient's EMR and will include telephone encounters, unscheduled clinic visits, ED visits, hospital admissions - total will be tallied.
Number of interviews/surveys completed | 2.5 years
  Patient and provider experience will be assessed with focus group discussions (FGDs), semi-structured interviews, and surveys

CONTACTS AND LOCATIONS:
Overall Officials: Brian Henick, MD, Principal Investigator — Assistant Professor of Medicine
Locations (4):
- United States (4):
  - Montefiore Health Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - NYU Medical Center, New York, New York
  - Columbia University Irving Medical Center, Herbert Irving Comprehensive Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hellmann MD, Paz-Ares L, Bernabe Caro R, Zurawski B, Kim SW, Carcereny Costa E, Park K, Alexandru A, Lupinacci L, de la Mora Jimenez E, Sakai H, Albert I, Vergnenegre A, Peters S, Syrigos K, Barlesi F, Reck M, Borghaei H, Brahmer JR, O'Byrne KJ, Geese WJ, Bhagavatheeswaran P, Rabindran SK, Kasinathan RS, Nathan FE, Ramalingam SS. Nivolumab plus Ipilimumab in Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2019 Nov 21;381(21):2020-2031. doi: 10.1056/NEJMoa1910231. Epub 2019 Sep 28. PMID 31562796
- [Background] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856
- [Background] Paz-Ares L, Ciuleanu TE, Cobo M, Schenker M, Zurawski B, Menezes J, Richardet E, Bennouna J, Felip E, Juan-Vidal O, Alexandru A, Sakai H, Lingua A, Salman P, Souquet PJ, De Marchi P, Martin C, Perol M, Scherpereel A, Lu S, John T, Carbone DP, Meadows-Shropshire S, Agrawal S, Oukessou A, Yan J, Reck M. First-line nivolumab plus ipilimumab combined with two cycles of chemotherapy in patients with non-small-cell lung cancer (CheckMate 9LA): an international, randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Feb;22(2):198-211. doi: 10.1016/S1470-2045(20)30641-0. Epub 2021 Jan 18. PMID 33476593
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Herbst RS, Baas P, Kim DW, Felip E, Perez-Gracia JL, Han JY, Molina J, Kim JH, Arvis CD, Ahn MJ, Majem M, Fidler MJ, de Castro G Jr, Garrido M, Lubiniecki GM, Shentu Y, Im E, Dolled-Filhart M, Garon EB. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. Lancet. 2016 Apr 9;387(10027):1540-1550. doi: 10.1016/S0140-6736(15)01281-7. Epub 2015 Dec 19. PMID 26712084
- [Background] Herbst RS, Giaccone G, de Marinis F, Reinmuth N, Vergnenegre A, Barrios CH, Morise M, Felip E, Andric Z, Geater S, Ozguroglu M, Zou W, Sandler A, Enquist I, Komatsubara K, Deng Y, Kuriki H, Wen X, McCleland M, Mocci S, Jassem J, Spigel DR. Atezolizumab for First-Line Treatment of PD-L1-Selected Patients with NSCLC. N Engl J Med. 2020 Oct 1;383(14):1328-1339. doi: 10.1056/NEJMoa1917346. PMID 32997907
- [Background] West H, McCleod M, Hussein M, Morabito A, Rittmeyer A, Conter HJ, Kopp HG, Daniel D, McCune S, Mekhail T, Zer A, Reinmuth N, Sadiq A, Sandler A, Lin W, Ochi Lohmann T, Archer V, Wang L, Kowanetz M, Cappuzzo F. Atezolizumab in combination with carboplatin plus nab-paclitaxel chemotherapy compared with chemotherapy alone as first-line treatment for metastatic non-squamous non-small-cell lung cancer (IMpower130): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2019 Jul;20(7):924-937. doi: 10.1016/S1470-2045(19)30167-6. Epub 2019 May 20. PMID 31122901
- [Background] Rittmeyer A, Barlesi F, Waterkamp D, Park K, Ciardiello F, von Pawel J, Gadgeel SM, Hida T, Kowalski DM, Dols MC, Cortinovis DL, Leach J, Polikoff J, Barrios C, Kabbinavar F, Frontera OA, De Marinis F, Turna H, Lee JS, Ballinger M, Kowanetz M, He P, Chen DS, Sandler A, Gandara DR; OAK Study Group. Atezolizumab versus docetaxel in patients with previously treated non-small-cell lung cancer (OAK): a phase 3, open-label, multicentre randomised controlled trial. Lancet. 2017 Jan 21;389(10066):255-265. doi: 10.1016/S0140-6736(16)32517-X. Epub 2016 Dec 13. PMID 27979383
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Almgren B, Lundqvist B, Eriksson I. [Local intra-arterial injection of reserpine in severe ischemia of the extremities--a good effect on ergotism]. Lakartidningen. 1984 Nov 7;81(45):4160-1. No abstract available. Swedish. PMID 6503493
- [Background] Beglarian AG, Arzumanian GA, Gevorkian LS. [Histochemical peculiarities of nucleoproteins in normal tissue, in foci of dyshormonal hyperplasia and in cancerous tumors of the breast]. Zh Eksp Klin Med. 1968;8(1):57-66. No abstract available. Russian. PMID 5761314
- [Background] Xing P, Zhang F, Wang G, Xu Y, Li C, Wang S, Guo Y, Cai S, Wang Y, Li J. Incidence rates of immune-related adverse events and their correlation with response in advanced solid tumours treated with NIVO or NIVO+IPI: a systematic review and meta-analysis. J Immunother Cancer. 2019 Dec 4;7(1):341. doi: 10.1186/s40425-019-0779-6. PMID 31801636
- [Background] Reynolds KL, Cohen JV, Ryan DP, Hochberg EP, Dougan M, Thomas M, Guidon A, Channick C, Chen ST, Schoenfeld S, Sise M, Leaf R, Neilan TG, Chu JN, Hur C, Murciano-Goroff Y, Villani AC, Nasrallah M, Sullivan RJ, Bardia A. Severe immune-related adverse effects (irAE) requiring hospital admission in patients treated with immune checkpoint inhibitors for advanced malignancy: Temporal trends and clinical significance. Journal of Clinical Oncology. 2018;36(15_suppl):3096-. doi: 10.1200/JCO.2018.36.15_suppl.3096.
- [Background] Zhou X, Yao Z, Yang H, Liang N, Zhang X, Zhang F. Are immune-related adverse events associated with the efficacy of immune checkpoint inhibitors in patients with cancer? A systematic review and meta-analysis. BMC Med. 2020 Apr 20;18(1):87. doi: 10.1186/s12916-020-01549-2. PMID 32306958
- [Background] Das S, Johnson DB. Immune-related adverse events and anti-tumor efficacy of immune checkpoint inhibitors. J Immunother Cancer. 2019 Nov 15;7(1):306. doi: 10.1186/s40425-019-0805-8. PMID 31730012
- [Background] de Zegher F, Jaeken J. Endocrinology of the carbohydrate-deficient glycoprotein syndrome type 1 from birth through adolescence. Pediatr Res. 1995 Apr;37(4 Pt 1):395-401. doi: 10.1203/00006450-199504000-00003. PMID 7596677
- [Background] Sun X, Roudi R, Dai T, Chen S, Fan B, Li H, Zhou Y, Zhou M, Zhu B, Yin C, Li B, Li X. Immune-related adverse events associated with programmed cell death protein-1 and programmed cell death ligand 1 inhibitors for non-small cell lung cancer: a PRISMA systematic review and meta-analysis. BMC Cancer. 2019 Jun 10;19(1):558. doi: 10.1186/s12885-019-5701-6. PMID 31182061
- [Background] Martins F, Sofiya L, Sykiotis GP, Lamine F, Maillard M, Fraga M, Shabafrouz K, Ribi C, Cairoli A, Guex-Crosier Y, Kuntzer T, Michielin O, Peters S, Coukos G, Spertini F, Thompson JA, Obeid M. Adverse effects of immune-checkpoint inhibitors: epidemiology, management and surveillance. Nat Rev Clin Oncol. 2019 Sep;16(9):563-580. doi: 10.1038/s41571-019-0218-0. PMID 31092901
- [Background] Osarogiagbon RU, Sineshaw HM, Unger JM, Acuna-Villaorduna A, Goel S. Immune-Based Cancer Treatment: Addressing Disparities in Access and Outcomes. Am Soc Clin Oncol Educ Book. 2021 Mar;41:1-13. doi: 10.1200/EDBK_323523. PMID 33830825
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Kotronoulas G, Kearney N, Maguire R, Harrow A, Di Domenico D, Croy S, MacGillivray S. What is the value of the routine use of patient-reported outcome measures toward improvement of patient outcomes, processes of care, and health service outcomes in cancer care? A systematic review of controlled trials. J Clin Oncol. 2014 May 10;32(14):1480-501. doi: 10.1200/JCO.2013.53.5948. Epub 2014 Apr 7. PMID 24711559
- [Background] Somerson NL, Ehrman L, Kocka JP. Induction by streptococcal L-forms of two reproductive isolating mechanisms in Drosophila paulistorum. Isr J Med Sci. 1984 Oct;20(10):1009-12. PMID 6439676
- [Background] US Department of Health and Human Services FaDA, Center for Drug Evaluation and Research, Center for Biologics Evaluation and Research, Center for Devices and Radiological Health. Guidance for industry: core patient-reported outcomes in cancer clinical trials. 2021 [cited 2021 6 August]. Available from: https://www.fda.gov/media/149994/download.
- [Background] Koot M, Keet IP, Vos AH, de Goede RE, Roos MT, Coutinho RA, Miedema F, Schellekens PT, Tersmette M. Prognostic value of HIV-1 syncytium-inducing phenotype for rate of CD4+ cell depletion and progression to AIDS. Ann Intern Med. 1993 May 1;118(9):681-8. doi: 10.7326/0003-4819-118-9-199305010-00004. PMID 8096374
- [Background] Sisodia RC, Rodriguez JA, Sequist TD. Digital disparities: lessons learned from a patient reported outcomes program during the COVID-19 pandemic. J Am Med Inform Assoc. 2021 Sep 18;28(10):2265-2268. doi: 10.1093/jamia/ocab138. PMID 34244760
- [Background] Gadgeel SM. Patient-Reported Outcomes in the Era of Immunotherapy Trials. J Thorac Oncol. 2021 Apr;16(4):516-518. doi: 10.1016/j.jtho.2021.02.014. No abstract available. PMID 33781441
- [Background] WhereWeLiveNYC. Explore Data- Where New Yokers Live 2018 [cited 2021 6 August]. Available from: https://wherewelive.cityofnewyork.us/explore-data/where-new-yorkers-live/.
- [Background] NYCHealth. Lung Cancer. 2021 [cited 2021 6 August]. Available from: https://www1.nyc.gov/site/doh/health/health-topics/lung-cancer.page.